CLINICAL TRIAL: NCT04007835
Title: Safety and Efficacy of Anlotinib Hydrochloride Combined With Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitors (EGFR TKIs) in Treating Advanced Non-small-cell Lung Cancer (NSCLC) Patients With Acquired Resistance to EGFR TKIs
Brief Title: Anlotinib Hydrochloride Combined With EGFR-Tyrosine Kinase Inhibitor (TKI) in Treating Advanced NSCLC Patients With Acquired Resistance to EGFR-TKI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangdong Association of Clinical Trials (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTONG1803
Record Dates: First submitted 2019-06-25; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: NSCLC
MeSH Terms: interventions — Gefitinib; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib Hydrochloride combined with EGFR-TKI (Experimental): Patients receive anlotinib (12 mg orally daily for 14 days every 21 days cycle) combined with one of following EGFR-TKIs: Gefitinib is administered 250 mg once per day. Erlotinib is administered 150 mg once per day , or Icotinib is administered 125 mg three times per day, until disease progression or untolerated toxicity.
  Interventions: Drug: Anlotinib Hydrochloride

INTERVENTIONS:
Drug: Anlotinib Hydrochloride — anlotinib (12 mg orally daily for 14 days every 21 days cycle) combined with one of EGFR-TKIs
  Other Names: Gefitinib Tablets; Erlotinib Hydrochloride Tablets; Icotinib Hydrochloride Tablets

SUMMARY:
The Single-arm, multicenter study evaluate the safety and efficacy of Anlotinib Hydrochloride combined with EGFR TKIs in treating Advanced NSCLC With acquired Resistance to EGFR TKIs

DETAILED DESCRIPTION:
EGFR TKI have been approved as first-line treatment in NSCLC patients harboring EGFR mutation. However, the acquired resistance of EGFR-TKI occurs almost constantly. Anlotinib is a novel oral multitarget tyrosine kinase inhibitor and primary targeted to Vascular Endothelial Growth Factor Receptor (VEGFR), fibroblast growth factor receptor (FGFR) , platelet-derived growth factor receptor (PDGFR) and c-Kit. The ALTER-0303 trial showed that patients with advanced non-small cell lung cancer (NSCLC) who received anlotinib as third-line or further therapy had more survival benefit. The Single-arm, multicenter study evaluate the safety and efficacy of Anlotinib Hydrochloride combined with EGFR TKIs in treating Advanced NSCLC With acquired Resistance to EGFR TKIs

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily participate in this study, signed and dated informed consent with good compliance and follow-up;
* Males or females aged 18 Years to 75 Years
* The patients should be confirmed with EGFR mutation [e.g., T 790 M , exon 19 deletion, L 858 R, etc],
* Cytologically or histologically confirmed locally advanced and / or metastatic non-small cell lung cancer (NSCLC).
* Patients should be using the EGFR TKI monotherapy as the first line treatment and meet the following criteria:

  1. Patients who showed objective clinical benefit from treatment with an EGFR

     TKI as defined by either:
     * Patients who showed complete (CR) or partial response (PR) ≥ 4 months, or
     * Patients who maintained stable disease (SD) status ≥ 6 months
  2. Patients who showed 1. risk of recurrence and progression, 2. gradual progression or local progression while on continuous treatment with EGFR TKI within the last 28 days prior to enrollment.( For recurrent diseases, patients can be accepted with adjuvant chemotherapy, neoadjuvant chemotherapy or neoadjuvant chemotherapy plus adjuvant chemotherapy in the past, and 3. relapse occurs 6 months after the end of treatment).

     1. CEA≥10ng/ml；
     2. Gradual progression: Disease control lasting ≥6 months with EGFR-TKI treatment, Compared with the previous assessment, no significant increment of tumor burden and progressive involvement of non-target lesions with a score less than 2, and Symptom scored ≤1. Local progression: Disease control lasting more than 3 months with EGFR-TKI treatment, Progressive disease (PD) due to solitary extracranial lesion or limitation in intracranial lesions (covered by a radiation field),and symptom scored ≤1
     3. Evidence of imaging or clinical progression is required if progression of disease occurs during the treatment or after the last treatment.
* At least one measurable lesion meet the requirements of the standard Response Evaluation Criteria In Solid Tumors（RESCIST）version 1.1
* Life expectancy is at least 3 months;
* Eastern Cooperative Oncology Group（ECOG）Performance Status（PS）:0-2.;
* The main organs function meet following criteria:

  * Blood routine examination criteria (no blood transfusion and blood products within 14 days, no correction by Granulocyte Colony-Stimulating Factor (G-CSF) and other hematopoietic stimuli): i) hemoglobin (HB) ≥90g/L ii) Absolute neutrophils count (ANC) ≥1.5×109/L iii) platelet (PLT) ≥80×109/L
  * Biochemical tests meet the following criteria i) total bilirubin (TBIL) ≤1.5 times of upper limit of normal (ULN); ii) alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤2.5 ULN, if liver metastasis occurred, ALT and AST ≤5 ULN; iii) serum creatinine (Cr) ≤1.25 ULN or creatinine clearance (CCr)≥45 mL/min
* Female patients of childbearing age agree that contraceptive measures must be used within the study period and within 8 weeks after the end of the study drug treatment. The serum or urine test indicates nonpregnant woman within 7 days prior to the study. Male patients agree to have contraceptive use during the study period and within 8 weeks after the end of the study period or have had surgical sterilization.

Exclusion Criteria:

* Small cell lung cancer (including Small cell lung cancer mixed with non-small cell lung cancer);
* Imaging (CT or MRI) showed that the distance between the lesion and the large vessels was less than 5 mm, or there were central tumors invading the local large vessels, or there were obvious pulmonary cavity or necrotic tumors.
* Patients with active brain metastasis, cancerous meningitis, spinal cord compression, or with brain or pia mater diseases detected by CT or MRI at screening time (patients with stable symptoms and complete treatment 14 days before enrollment may be admitted to the group, but no symptoms of cerebral hemorrhage should be confirmed by craniocerebral MRI, CT or venography evaluation).
* Uncontrollable hypertension (systolic blood pressure ≥ 140 mmHg, or diastolic blood pressure ≥ 90 mmHg, despite using the optimal medical treatment;
* Patients are participating in other clinical studies, or there are less than four weeks before the end of the previous clinical study.
* Other active malignant tumors requiring concurrent treatment;
* The patient has a history of malignant tumors. Patients with basal cell carcinoma of skin, superficial bladder cancer, squamous cell carcinoma of skin or carcinoma of cervix in situ who had undergone possible curative treatment and had no disease recurrence within 5 years after the initiation of curative treatment are permitted.
* Patients had treatment related adverse reactions after previous systemic anti-tumour therapy (except hair loss), but did not recover to NCI-CTCAE ≤ 1 grade.
* The patient has the coagulation disorders (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or activated partial thromboplastin time (APTT) > 1.5 ULN), or bleeding tendency, or undergoing thrombolysis or anticoagulation therapy; Note: On the premise that the International Standardized Ratio of Prothrombin Time (INR) is less than 1.5, low doses of heparin (0.6 million to 12,000 U per day for adults) or aspirin (less than 100 mg per day) are allowed for preventive purposes.
* Renal insufficiency: Urinary routine indicated that urinary protein ≥ ++ or confirmed 24-hour urinary protein ≥ 1.0 g;
* Subjects who had undergone major surgery or had severe trauma had less than 14 days before enrollment.
* Severe acute or chronic infections requiring systemic treatment
* Severe cardiovascular diseases: grade II or above myocardial ischemia or myocardial infarction and poor control arrhythmias (including corrected QT interval (QTc) interval ≥ 450 ms for males and ≥ 470 ms for females); cardiac insufficiency of grade III to IV according to New York Heart Association (NYHA) criteria, or left ventricular ejection fraction (LVEF) < 50% by color Doppler echocardiography;
* ≥ CTCAE grade 2 peripheral neuropathy, except for trauma.
* Respiratory syndrome (≥ CTCAE grade 2 dyspnea), serous effusion (including pleural effusion, ascites, pericardial effusion) requiring surgical treatment;
* Long-term unhealed wound or fracture;
* Decompensated diabetes mellitus or other contraindications of high-dose glucocorticoid therapy;
* There are obvious factors affecting oral drug absorption, such as inability to swallow, chronic diarrhea and intestinal obstruction;
* Three months prior to enrollment, significant hemoptysis (more than 50 ml per day) occurred, or significant clinical hemorrhage symptoms or defined bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood ++ or above, or suffering from vasculitis.
* Arteriovenous thrombosis events occurred within 12 months before enrollment, such as cerebrovascular accident (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism.
* Patients participated in clinical trials of other antineoplastic drugs within four weeks prior to enrollment, or planned systemic anti-tumor therapy within four weeks prior to enrollment or during the period of the study, including cytotoxic therapy, signal transduction inhibitors, immunotherapy (or use of mitomycin C within six weeks prior to the treatment of the experimental drugs). Over-extended-field radiotherapy (EF-RT) was performed within four weeks prior to grouping or limited-field radiotherapy to evaluate the tumor lesions was performed within two weeks prior to grouping;
* Physical and laboratory findings Untreated active hepatitis (hepatitis B: HBsAg positive and hepatitis B virus (HBV) DNA ≥ 500 IU/mL; hepatitis C: hepatitis C virus (HCV) RNA positive and abnormal liver function); co-infection of hepatitis B and hepatitis C;
* According to the researcher's judgment, patients may have other factors that may lead to the forced termination of the study, such as other serious diseases or serious abnormal laboratory examinations or other factors that may affect the safety of the subjects, or family or social factors such as test data and sample collection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival（PFS） | From randomization to the first occurrence of disease progression or death from any cause, whichever occurs earlier, assessed up to 1 year

SECONDARY OUTCOMES:
6 months and 12 months progression-free survival (PFS) Rate | Up to 1 year
objective response rate (ORR) | Up to 1 year
Disease Control Rate(DCR) | Up to 1 year
Overall survival (OS) | From the date of randomization to the date of death from any cause，assessed up to 2 year
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 21 days post-the last treatment
  Adverse Events
progression-free survival (PFS) for different types of EGFR mutation | Up to 1 year
Overall survival (OS) for different types of EGFR mutation | Up to 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Long Wu, MD, Study Chair — Guangdong General Hospital (GGH)& Guangdong Academy of Medical Sciences; HUAJUN CHEN, MD, Study Director — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Chen HJ, Tu HY, Hu Y, Fan Y, Wu G, Cang S, Yang Y, Yang N, Ma R, Jin G, Xu X, Liu A, Tang S, Cheng Y, Yu Y, Xu CR, Zhou Q, Wu YL. A phase II trial of anlotinib plus EGFR-TKIs in advanced non-small cell lung cancer with gradual, oligo, or potential progression after EGFR-TKIs treatment (CTONG-1803/ALTER-L001). J Hematol Oncol. 2025 Jan 5;18(1):3. doi: 10.1186/s13045-024-01656-0. PMID 39757186